CLINICAL TRIAL: NCT06476496
Title: Pain Relief With Integrative Medicine (PRIMe)?: Feasibility of Acupuncture for Long COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Nikki Gentile, Assistant Professor, Family Medicine, University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00019169; R34AT012679-01 (NIH)
Record Dates: First submitted 2024-06-24; First posted 2024-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Long COVID; Pain
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture (Experimental): Participants will receive 8 sessions of acupuncture treatment
  Interventions: Procedure: Acupuncture
- Usual Care (No Intervention): Participants will continue to receive any current or recommended treatments from their doctors for their long COVID symptoms.

INTERVENTIONS:
Procedure: Acupuncture — A licensed acupuncturist will insert sterile disposable acupuncture needles in the selected body and ear acupoints aiming to alleviate long COVID related pain symptoms. Needles will be removed after 20 minutes of retention. After all the needles are removed, the acupuncturist will insert Pyonex press tack needles (0.3mm) in the participants' left ears and suggest the participants retain them in their ears for up to 5 days.
  Arms: Acupuncture

SUMMARY:
The goal of this preliminary study is to test methods and procedures to be used in a fully-powered trial to evaluate acupuncture treatment effectiveness. Specifically, we will test the feasibility of conducting a 2-arm randomized clinical trial for evaluating the effectiveness of acupuncture for pain in patients with long COVID. Researchers will compare pain intensity and impact on general activities over 5 months in those who receive acupuncture treatment compared to patients who are receiving usual long COVID care.

Participants will complete 4 online surveys at weeks 0, 4, 8, and 20. These surveys include validated mental and physical health questionnaires. Participants who are randomly selected to receive the intervention will receive 8 acupuncture treatment sessions.

DETAILED DESCRIPTION:
Long-COVID has negatively impacted millions of individuals' quality of life, daily functioning, and ability to work, and has placed enormous demands on the healthcare system. Pain-related symptoms are reported by a large subset of patients with long COVID, and yet pain is still not consistently addressed in workups or treatment plans. Thus, we have chosen to study acupuncture for improving pain, quality of life, and function in individuals experiencing long COVID-related pain. Acupuncture has been shown to be successful in treating various types of chronic pain and should lend itself to similar results with pain related to long COVID. Furthermore, acupuncture focuses on treating the whole patient, which makes it uniquely well-suited for a complex condition affecting multiple body systems, like long COVID.

We propose an initial study to determine the feasibility of successfully conducting a subsequent fully-powered pragmatic randomized trial evaluating the effectiveness of Traditional Chinese Medicine (TCM) acupuncture for persistent pain problems experienced by persons with long COVID. Acupuncture is a physical treatment that aims to correct imbalances in the body (including inflammation and pain) within a Chinese Medicine paradigm.

Our specific aims are to:

1. Assess the feasibility of conducting a randomized clinical trial comparing acupuncture with usual care alone for reducing pain in patients with long COVID;
2. Evaluate the overall patient experience with participation in the feasibility trial and solicit suggestions about how the study procedures, documents, and treatment protocols could be improved to facilitate participation and better meet participants' needs; and
3. Revise study procedures, protocols, and instruments to prepare for a fully-powered pragmatic randomized trial.

Participants randomized to acupuncture will receive a total of 8 weekly individual treatments lasting one hour each. Participants will lie supine on a treatment table while the acupuncturist inserts needles in selected body points. Bilateral needling of the pre-specified acupuncture points will be performed according to TCM principles and will include efforts to obtain De Qi.

This study has the potential to help patients with long COVID improve function and quality of life, and to provide clinicians with more tools to effectively respond to their patients' needs. This study will occur through the University of Washington (UW) Long COVID Clinic at the UW Primary Care Northgate Clinic site.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at the time of consent.
* Previous suspected, probable, or confirmed SARS-CoV-2 infection, as defined by the Pan American Health Organization
* Report pain symptoms including musculoskeletal pain (joint, muscle, bone pain), chest pain, abdominal pain, headache, back pain, nerve pain, and pain in ear following a SARS-CoV-2 infection that has persisted for at least 12 weeks and is still present at the time of consent.
* Report pain intensity (0-10 scale) ≥4 in the last 7 days.28
* As of today, has been seen by a clinician in the UW Long COVID Clinic either in-person or via telehealth/virtual visit
* Able to speak and read English and provide informed consent to complete the study requirements.

Exclusion Criteria:

* <18 years of age at the time of consent.
* Reports absence of pain, pain for less than 12 weeks, or a pain intensity <4 over the last 7 days.
* Report baseline level of pain for those who have pre-existing chronic pain (i.e., chronic pain condition(s) present prior to COVID-19 illness AND chronic pain not worsened post-COVID).
* Already received acupuncture treatment for long COVID symptoms.
* Unable to travel to the UW Northgate Clinic once a week for 8 weeks for acupuncture treatments.
* Has seizure disorder with high risk of seizure (i.e., new diagnosis of seizure disorder and/or new medication in the last 3 months, or uncontrolled/unclear triggers for seizures).
* Is currently Pregnant
* Is receiving active cancer therapy
* Has severe neutropenia (<500 WBC) due to any cause within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Pain, Enjoyment and General Activity (PEG) | Weeks 0, 4, 8, 20
  A pain-related predictor is an easily-understood three-question instrument that asks about average pain, enjoyment of life, and general activity in the past week on a 0 to 10 scale.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale (PCS) | Weeks 0, 8, 20
  A self-report measure of catastrophic thinking related to pain, including subscales of rumination, magnification, and helplessness.
PROMIS-29 | Weeks 0, 8, 20
  A questionnaire covering 7 domains (anxiety, sleep, depression, physical function, pain intensity, social roles, and fatigue) of mental and physical health.
PROMIS Cognitive Function | Weeks 0, 8, 20
  Assesses patient-perceived cognitive deficits. Facets include mental acuity, concentration, verbal and nonverbal memory, verbal fluency, and perceived changes in cognitive functions.
UW Pain Related Self-Efficacy Scale (PRSE) | Weeks 0, 8, 20
  A measure self-efficacy. Expectation for recovery is measured using an 11-point numerical rating scale (0=no confidence in recovery, 10=complete confidence in recovery) using the question: "How confident are you that your pain will be completely gone or much better 3 months from now?"

CONTACTS AND LOCATIONS:
Overall Officials: Nikki Gentile, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- UW Medicine Primary Care at Northgate, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No